CLINICAL TRIAL: NCT05906719
Title: Machine Vision Based Machine Rating of MDS-UPDRS III
Brief Title: Machine Vision Based MDS-UPDRS III Machine Rating
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Second Affiliated Hospital of Soochow University (Other); Beijing Hospital (Other Government); Beijing Tiantan Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Fujian Medical University Union Hospital (Other); Guangdong Provincial People's Hospital (Other); West China Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: u3
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-03

CONDITIONS: Parkinsonian Disorders; Machine Learning
MeSH Terms: conditions — Parkinsonian Disorders | interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: video recording — Patients' performance of MDS-UPDRS III will be recorded.

SUMMARY:
The Movement Disorders Society (MDS) Unified Parkinson's Disease Rating Scale (UPDRS) Part III (MDS-UPDRS III) is the primary assessment method for motor symptoms in Parkinson's disease patients. Currently, movement disorder specialists conduct semi-quantitative scoring, which entails limitations such as subjectivity, weak sensitivity, and a limited number of professional physicians. This study, based on machine vision, establishes gold standard labels according to expert scoring. By using machine learning, we develop a machine rating model and compare the model's performance with gold standard rating and general clinical rating to investigate the accuracy of machine vision-based MDS-UPDRS III machine rating.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for Parkinsonism established by the International Movement Disorder Society: having bradykinesia, and meeting at least one of the two criteria for resting tremor or muscle rigidity
* 20 to 80 years old
* Good compliance, voluntarily joining the study, and able to sign an informed consent form or have it signed by a legal representative

Exclusion Criteria:

* Significant cognitive impairment (MMSE ≤ 23)
* Unable to sign written informed consent or unable to complete the trial due to other reasons
* Other situations in which the researcher deems the participant unsuitable for this study
* Participation in other clinical trials

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, participants are mainly recruited from the Department of Neurology at Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, as well as from movement disorder clinics at 7 other centers. Participants are enrolled through outpatient assessment and screening. Two specialists in movement disorders independently diagnosed participants as having "Parkinsonism". In cases where there is a diagnostic disagreement, the Movement Disorder Specialist Group at the Department of Neurology, Ruijin Hospital collectively discusses and makes the decision.
Sampling Method: Probability Sample
Enrollment: 871 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
ACC0 of machine rating vs gold standard rating | 1 day
  The accuracy rate when machine rating equals gold standard rating.
ACC1 of machine rating vs gold standard rating | 1 day
  The accuracy rate when machine rating equals the range of gold standard rating plus or minus one.
Weighted kappa of machine rating vs gold standard rating | 1 day
  The weighted kappa when machine rating equals gold standard rating.
Lin's CCC of machine rating vs gold standard rating | 1 day
  The Lin's Concordance Correlation Coefficient when machine rating equals gold standard rating.

SECONDARY OUTCOMES:
Accuracy rate of machine rating vs general clinical rating | 1 day
  Comparing the absolute residuals between machine rating and the gold standard rating with the absolute residuals between general clinical raitng and the gold standard rating.
Accuracy rate of machine facilitated rating vs general clinical rating | 1 day
  Comparing the absolute residuals between machine facilitated rating and the gold standard rating with the absolute residuals between general clinical raitng and the gold standard rating.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Center for Movement Disorders, Department of Neurology, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Neurology Department, Beijing, Beijing Municipality
  - Department of Neurology, Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Department of Neurology, Guangdong Neuroscience Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong
  - Department of Neurology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Department of Neurology and Clinical Research Center of Neurological Disease, The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Department of Neurology and Institute of Neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Neurology, West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No